CLINICAL TRIAL: NCT02588976
Title: Evaluation of a New Sonoclot Device for Heparin Management in Cardiac Surgery
Acronym: SONEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Triemli Hospital (Other)
Responsible Party: Principal Investigator, Christoph K Hofer, Prof. Dr. med, Triemli Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STZ-Dendrite06
Record Dates: First submitted 2015-10-23; First posted 2015-10-28 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Diagnostic Techniques and Procedures; Cardiac Surgical Procedure
Keywords: Activated clotting time; Sonoclot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACT measurements (Other): ACT measurements by SONOCLOT Analyzer during cardiac surgery
  Interventions: Device: Sonoclot Analyzer

INTERVENTIONS:
Device: Sonoclot Analyzer — Blood coagulation test during cardiac surgery: Measurement of activated clotting time during cardiac surgery by Sonoclot Analyzer

SUMMARY:
The SONOCLOT Analyzer (S1; Sienco, Inc. Boulder, CO USA, Model DP-2951) is used to perform kaolin-based activated clotting time as routine monitor of heparin therapy in patients undergoing cardiac operations. In addition, the device allows the assessment of the patient's coagulation status by a glass-bead activated test. Recently, a new SONOCLOT analyzer (S2) has been developed. As part of the routine management using S1, tests are also performed on S2. Results are entered into the cardiac surgery data base of all cardiac surgery patients and analyzed.

DETAILED DESCRIPTION:
The SONOCLOT Analyzer (S1; Sienco, Inc. Boulder, CO USA, Model DP-2951) is used to routinely perform kaolin-based activated clotting time (kACT) as monitor of heparin therapy in patients undergoing cardiac operations on cardiopulmonary bypass.

Apart from kACT, the device allows the assessment of the patient's coagulation status by a glass-bead activated test (gbACT+, depicting also clot rate = CR and platelet function = PF). Recently, a new SONOCLOT analyzer (S2) has been developed. Although the S2 shares the technical fundamentals with the S1, the redesign of the device may result in performance changes of kACT and gbACT.

Routine management in cardiac surgery patients is guided using S1 and addition, tests are run on S2. Data are entered into the the cardiac surgery data base and S1 and S2 performance is compared by Bland-Altman analysis and % error calculation in order to establish new reference values.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive cardiac surgery patients

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Genoni, MD, Study Chair — Triemli City Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganter MT, Hofer CK. Coagulation monitoring: current techniques and clinical use of viscoelastic point-of-care coagulation devices. Anesth Analg. 2008 May;106(5):1366-75. doi: 10.1213/ane.0b013e318168b367. PMID 18420846

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACT Measurements
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 30

OUTCOME MEASURES:

1. Primary Outcome: Kaolin-activated Clotting Time
Time Frame: Routine measurements during cardiac surgery
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | All Patients
Number analyzed (Participants) | 30
seconds | 309 (211)

2. Secondary Outcome: Glass Bead Activated Clotting Time
Time Frame: Routine measurements during cardiac surgery
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | ACT Measurements
Number analyzed (Participants) | 30
seconds | 195 (57)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No